CLINICAL TRIAL: NCT01423201
Title: TIA Triage Trial and Evaluation of Vascular-Specific Inflammatory BiomarkerLp-PLA2 as a Stratification Tool for TIA Triage and Stroke Risk
Brief Title: Transient Ischemic Attack (TIA) Triage and Evaluation of Stroke Risk
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Diadexus, Inc. (Industry); University of California, Davis (Other)
Responsible Party: Principal Investigator, Gregory W Albers, MD, Professor of Neurology, Stanford University
Other Study IDs: SU-08012011-8167; 19211
Record Dates: First submitted 2011-08-16; First posted 2011-08-25 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Cerebrovascular Accident
Keywords: TIA; triage; Lp-PLA2; Proteomic; Genomic
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — First 100 cases:
  2 tiger top or gold top tubes 2 lavender top tubes
  * Blood specimens should be inverted 10 times before processing.
  * Centrifuge and separate within four hours of venipuncture.
  * Transfer 1.0 ml into 2 transfer tubes
  Freeze at -70 C
  Additional 80 cases:
  3 PAXgene tubes (total 16cc) - containing 7.5 cc preservative to stabilize RNA immediately.
  Invert 20 times then sit at room temperature overnight Place into a -70C freezer until processed
  2 tiger top or gold top tubes 2 lavender top tubes
  * Blood specimens should be inverted 10 times before processing.
  * Centrifuge and separate within four hours of venipuncture.
  * Transfer 1.0 ml into 2 transfer tubes
  Freeze at -70 C
Oversight: Data Monitoring Committee: No

SUMMARY:
Transient ischemic attack (TIA) is a transient neurological deficit (speech disturbance, weakness…), caused by temporary occlusion of a brain vessel by a blood clot that leaves no lasting effect.

TIA diagnosis can be challenging and an expert stroke evaluation combined with magnetic resonance imaging (MRI) could improve the diagnosis accuracy.

The risk of a debilitating stroke can be as high as 5% during the first 72 hrs after TIA.

TIA characteristics (duration, type of symptoms, age of the patient), the presence of a significant narrowing of the neck vessels responsible for the patient's symptoms (symptomatic stenosis), and an abnormal MRI are associated with an increased risk of stroke.

An emergent evaluation and treatment of TIA patients by a stroke specialist could reduce the risk of stroke to 2%.

Stanford has implemented an expedited triage pathway for TIA patients combining a clinical evaluation by a stroke neurologist, an acute MRI of the brain and the vessels and a sampling of biomarkers (Lp-PLA2). The investigators are investigating the yield of this unique approach to improve TIA diagnosis, prognosis and secondary stroke prevention. The objective of this prospective cohort study is to determine which factors will help the physician to confirm the diagnosis of TIA and to define the risk of stroke after a TIA.

DETAILED DESCRIPTION:
Patients with a clinical suspicion of TIA seen at the Stanford Emergency Department, will be admitted to the Clinical Decision Area (CDA). The CDA is a short duration (<24 hrs)) hospitalization unit, where the patient can receive expedited evaluation and monitoring in a more comfortable setting than in the ED. Patients will be evaluated by a neurologist (resident with fellow or stroke attending). Clinical information will be collected in a dedicated chart.

Evaluation:

As recommended by the AHA, in the absence of contraindications, all the patients will undergo an MRI of the brain and a neck vessel evaluation as part of standard care. This exam will be obtained within 6 hours after patient admission to the emergency department. The diffusion sequence of the brain MRI will detect the presence of an acute injury related to a blood clot (ischemic injury), and the perfusion sequence will capture abnormal intra-cerebral blood flow. The other sequences will exclude the presence of other brain lesions susceptible to explain the transient symptoms presented by the patient. The MR angiogram (MRA) of the neck and intracranial vessels will detect the presence of a symptomatic stenosis that would require emergent treatment. In case of MRI contraindication, the patient will undergo a CT of the head and neck combining neck and intracranial vessel evaluation and perfusion imaging.

As recommended, patients will get an EKG and a cardiovascular examination as part of routine care.

As recommended, patients will get a standard lab evaluation as part of routine care including general chemistry, hematology, coagulation, lipid profile, Hb A1C), and if indicated, a specific prothrombotic and an inflammatory evaluation.

In approximately 100 patients - AS PART OF THIS RESEARCH PROTOCOL - the investigators will evaluate the level of the lipoprotein A2 L at one time point. This biomarker has been associated in one publication with an increased risk of vascular events among TIA patients. After informed consent, the investigators will perform a standard venipuncture to draw 10 mL of blood per patient. The blood will be collected in serum gel separator tubes. The serum will be kept cold, and separated from gel and cells within 2 hours. The specimens will then be frozen down at -70C until analyses performed by diaDexus lab who are sponsoring this part of the study.

* As part of the routine triage pathway, patients with an initial normal clinical, radiological and biological evaluation are evaluated within the next 12 hours by an attending stroke neurologist who will determine whether the patient could be safely discharged from the hospital, and the treatment plan including risk factors management and antithrombotic treatment. This treatment is initiated in the hospital before patient discharge. In following these guidelines, the majority of patients are hospitalized for less than 24 hours.
* As part of the routine triage pathway, all patients are seen by a stroke neurologist and/or a stroke trained nurse practitioner within the next 2 weeks at the Stanford outpatient TIA clinic. All the patients routinely receive a follow up telephone call at 1 month, 3 months and 1 year to evaluate the occurrence of a stroke a myocardial infarction and/or a vascular death. In some instances, one or more of these visits is clinically indicated to be an in-person visit. If this is the case, the data from the in-person clinic visit will be used as part of this study rather than a telephone visit.

The clinical characteristics of the TIA, the radiological results, the biological results and the follow up information will be collected and used in this research protocol for all the consented patients.

The investigators will include all patients who were evaluated under this new pathway since it's inception in January 2010. This patient population will be included as chart reviews. The charts will be reviewed and data points extracted from the medical record to be used as part of the research.

An additional arm was added in 2012:

A biomarker of ischemia may help the physicians to confirm the diagnosis of TIA, and help to stratify the risk among patients with negative brain imaging. Researchers at UC Davis, have evaluated gene expression profiles after a stroke in circulating leucocytes. They have isolated specific gene expression profiles associated with transient brain ischemia. The aim of this study is to define whether gene expression and proteomic profiles may help to detect ischemic mechanism of transient neurological symptoms and stratify the risk of future stroke in patients with a negative MRI.

We will prospectively collect blood samples at Stanford University and the samples will be shipped to UC Davis for processing and interpretation.

Patients: 80 patients at Stanford evaluated for suspicion of TIA with a discharge diagnosis of ischemic event: Transient Ischemic Attack or Brain Infarction with transient or minor neurological symptoms (NIHSS≤2).

Blood Tests:

Genomic analyses: we will evaluate the whole blood genomic profiles. Blood will be collected into 3 PAXgene tubes (total 16cc). The FDA approved tubes contain 7.5 cc preservative to stabilize RNA immediately. The tubes will be inverted 20 times sit at room temperature overnight then placed into a -70C freezer until processed. Those samples will be sent to be processed by Professor Frank Sharp's Lab at UC Davis. The RNA will be processed using Affymetrix whole genome arrays. In addition, blood is drawn into a lavender top and tiger top tubes, processed and stored at Stanford University for future research studies.

Proteomic analyses will be performed on standard serum tubes as mentioned above. Proteomics analyses will be processed and interpreted in collaboration with Dr. Frank Sharp's group.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women age greater than 18 year old
* Symptoms suggestive of an acute TIA

Exclusion Criteria:

* Patients with contraindication to brain imaging: MRI and CT.
* Patient with persistent major deficit (NIHSS> or = 4)
* Informed consent could not be obtained either directly from the patient or from legally authorized representative.
* Severe coexisting or terminal systemic disease with like expectancy below 90 days or that may interfere with the conduct of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the ED with symptoms of acute TIA
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2010-09; Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
vascular events | 90 days

SECONDARY OUTCOMES:
Vascular Events | 7 days
Vascular Events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gregory W Albers, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - UC Davis Medical Center, Davis, California
  - Stanford University School of Medicine, Stanford, California
  - Michigan State University, Grand Rapids, Michigan

REFERENCES:
- [Background] Easton JD, Saver JL, Albers GW, Alberts MJ, Chaturvedi S, Feldmann E, Hatsukami TS, Higashida RT, Johnston SC, Kidwell CS, Lutsep HL, Miller E, Sacco RL; American Heart Association; American Stroke Association Stroke Council; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; Interdisciplinary Council on Peripheral Vascular Disease. Definition and evaluation of transient ischemic attack: a scientific statement for healthcare professionals from the American Heart Association/American Stroke Association Stroke Council; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; and the Interdisciplinary Council on Peripheral Vascular Disease. The American Academy of Neurology affirms the value of this statement as an educational tool for neurologists. Stroke. 2009 Jun;40(6):2276-93. doi: 10.1161/STROKEAHA.108.192218. Epub 2009 May 7. PMID 19423857
- [Background] Cucchiara BL, Messe SR, Sansing L, MacKenzie L, Taylor RA, Pacelli J, Shah Q, Kasner SE. Lipoprotein-associated phospholipase A2 and C-reactive protein for risk-stratification of patients with TIA. Stroke. 2009 Jul;40(7):2332-6. doi: 10.1161/STROKEAHA.109.553545. Epub 2009 May 21. PMID 19461040